CLINICAL TRIAL: NCT04151589
Title: Work Flow Improvement in Pre-procedural Management of Acute Ischemic Stroke With Endovascular Treatment: a Multi-centre, Cluster Randomised, Open Label, Parallel Controlled Study
Brief Title: Endovascular Treatment Key Technique and Emergency Work Flow Improvement of Acute Ischemic Stroke (ANGEL-ACT): Phase Two
Acronym: ANGEL-ACT II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director of Department of interventional neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016YFC1301501-2
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Intracranial Artery Occlusion With Infarction (Disorder)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Site (Experimental): The process below will be allocated in Interventional Sites:
  1. At each interventional sites, implementing full assessment of current emergency work flow of acute ischemic stroke patients who eligible for endovascular treatment. All interventional sites would undergo assessment in order to form a baseline.
  2. Drafting intervention approaches based on the assessment results of all interventional sites. These approaches are executable, reproducible, and measurable.
  3. Emergency work flow management APP would be installed on smartphones of designated personnel at each interventional sites.
  4. Both intervention approaches and APP would be incorporated with original work flow at each interventional site.
  5. Training sessions would be held in interventional sites or online every 3 month once the patient enrolment begin.
  6. Outcome data would be analysed and dispatched every 3 month for each interventional sites.
  Interventions: Behavioral: ANGEL Intervention Package and Toolbox
- Control Site (No Intervention): The control site would not undergo any emergency work flow modification for acute ischemic stroke patients who eligible for endovascular treatment.

INTERVENTIONS:
Behavioral: ANGEL Intervention Package and Toolbox — The interventional measures include emergency work flow management app on smartphone, specialized training, assessment of quality improvement outcomes and feedback on a regular basis, patient-centred management frame based lean six-sigma, and other specialised approach.
  Arms: Interventional Site

SUMMARY:
The study is the second phase of Endovascular Treatment Key Technique and Emergency Work Flow Improvement of Acute Ischemic Stroke (ANGEL-ACT).

During the first phase of the ANGEL-ACT (NCT03370939, a prospective multi-center registry study), problems and difficulties in the emergency work flow of acute ischemic stroke care in China have been identified, such as inadequate pre-hospital notification, delay of in-hospital diagnosis and treatment, difficulty in treatment consent, lack of professional training of endovascular treatment,etc., especially in the delay of in-hospital diagnosis and treatment.

ANGEL-ACT II is a cluster randomized, parallel controlled study. The aim of this study was to evaluate the effectiveness of multi-modal medical quality improvement measures on the delay of hospital-level emergency work flow of acute ischemic stroke management as well as its impact on patient prognosis. The interventional measures include emergency work flow management app on smartphone, specialized training, assessment of quality improvement outcomes and feedback on a regular basis.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, cluster randomized, open label, parallel controlled study that enrolled patients with acute ischemic stroke who underwent endovascular treatment in about 34 hospitals in China. The ratio Interventional arm control arm is 1:1, which means 17 hospitals and 332 participants in each arm.

ELIGIBILITY:
Investigational Sites Inclusion Criteria:

* Participated in the ANGEL-ACT registry study
* Secondary or tertiary hospitals
* Available of emergency department and neurology ward for stroke patients
* Must have 24 hours × 7 days emergency department for stroke
* Capable of rt-PA thrombolysis and endovascular treatment

Investigational Sites Exclusion Criteria

* Endovascular treatment volume < 20 per year
* Unwillingness to participate ANGEL-ACT II and follow the protocol
* Currently participating other stroke treatment improving program/project or similar clinical studies

Participant Inclusion Criteria

* Age ≥ 18 years old
* Admitted from emergency or outpatient department;
* Acue ischemic stroke with large artery occlusion
* Within 24 hours after the onset, and eligible for endovascular treatment.
* The patient or legal representative give written informed consent

Participant Exclusion Criteria:

* Unsuitable for this study investigators' discretion
* Progressive stroke or in-hospital stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of reaching the standard arrival-to-groin Puncture time | From the time of arrival at the emergency department until the time of successful groin puncture, assessed up to 12 hours
  The percentage of reaching the guideline recommended time target for acute ischemic stroke patients who eligible for endovascular treatment.

SECONDARY OUTCOMES:
Time from arrival to groin puncture | From the time of arrival at the emergency department until the time of successful groin puncture, assessed up to 12 hours
  Minutes
Time from arrival to imaging | From the time of arrival at the emergency department until the time of brain imaging, assessed up to 12 hours
  Minutes
Time from imaging to groin puncture | From the time of brain imaging until the time of successful groin puncture, assessed up to 12 hours
  Minutes
Time from groin puncture to recanalization | From the time of successful groin puncture until the time of the recanalization of the occluded artery, assessed up to 4 hours
  Minutes
Time from arrival to recanalization | From the time of arrival at the emergency department until the time of the recanalization of the occluded artery, assessed up to 48 hours
  Minutes
Time from symptom onset to recanalization | From the time of symptom onset until the time of of the recanalization of the occluded artery, assessed up to 48 hours
  Minutes
Recanalization rate immediately after the procedure | Immediately after the procedure
  modified thrombolysis in cerebral infarction (mTICI) 2b-3
Recanalization rate 24 hours after the procedure | 24 hours after the procedure
  Recanalization was defined as a thrombolysis in myocardial infarction (TIMI ) score of 2- 3.
Modified Rankin Scale independence rate within 90 days after the procedure | 90 days after enrolment
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. (Score Description: 0---No symptoms at all. 1---No significant disability despite symptoms; able to carry out all usual duties and activities. 2---Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3---Moderate disability; requiring some help, but able to walk without assistance. 4--- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5---Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6---Dead. In clinical practice, mRS ≤ 2 means good outcome. Modified Rankin Scale independence rate refers to the percentage of participants with mRS less than 3 after treatment.
EQ-5D-3L 90 days after the procedure | 90 days after the procedure
  The EQ-5D-3L essentially consists of two pages: the EQ-5D descriptive system and the EQ-5D visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems (labelled 1-3). The respondent is asked to indicate his / her health state by checking the box against the most appropriate statement in each of the five dimensions. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine'( score as 100) and 'The worst health you can imagine' (score as 0). This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Rate of symptomatic intracerebral hemorrhage within 24 hours after the procedure | 24 hours within the procedure ended
Rate of complications related to the procedure | 24 hours after the procedure
Rate of all cause mortality within 90 days after the procedure | 90 days after enrolment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided